CLINICAL TRIAL: NCT06899139
Title: Myopia Adjustment Using Dual-intervention: Red-Light Therapy & Innovative Design in Orthokeratology
Acronym: MADRID
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Miopía Fernández-Velázquez (Network)
Responsible Party: Principal Investigator, Fernando Fernandez Velazquez, Doctor of Optometry, Centro de Miopía Fernández-Velázquez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMFV-SCL-2024-04
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: MYOPIA
Keywords: Myopia; Orthokeratology; Red-Light Therapy; RLRL
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group randomized controlled trial. Participants will be allocated in a 1:1 ratio to either the experimental group (Orthokeratology + Repeated Low-Level Red-Light Therapy) or the control group (Orthokeratology only). Randomization will be computer-generated and stratified to ensure balanced group sizes. The intervention will be applied continuously for 6 months, with a possible extension to 12 months based on interim evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm Title: Orthokeratology + Red-Light Therapy Control Arm Title: Orthokeratology Only (Experimental): 1st Experimental Arm: Orthokeratology + Red-Light Therapy Participants in this arm will wear orthokeratology (OK) lenses overnight for at least 8 hours per night and undergo repeated low-level red-light (R.L.R.L.) therapy twice daily. Each R.L.R.L. session will last up to 3 minutes, with a minimum interval of 4 hours between sessions. The intervention period will last 6 months, with a potential extension to 12 months based on clinical assessment.
  Interventions: Device: Repeated Low-Level Red-Light Therapy Intervention Type: Device Description: Participants in the experimental group will receive repeated low-level red-light (R.L.R.L.) therapy twice daily using a no
- 2nd Control Arm: Orthokeratology Only (Active Comparator): Participants in this arm will wear orthokeratology (OK) lenses overnight for at least 8 hours per night. They will not receive red-light therapy. The intervention period will last 6 months, with a potential extension to 12 months based on clinical assessment.
  Interventions: Other: Orthokeratology Lens Wear

INTERVENTIONS:
Other: Orthokeratology Lens Wear — Orthokeratology Lens Wear
  Intervention Type:
  Device
  Description:
  Participants will wear gas-permeable orthokeratology (OK) lenses overnight for a minimum of 8 hours per night. Lenses are designed to reshape the cornea temporarily to reduce refractive error and slow axial elongation. This intervention is administered to both the experimental and control groups.
  Arms: 2nd Control Arm: Orthokeratology Only
Device: Repeated Low-Level Red-Light Therapy Intervention Type: Device Description: Participants in the experimental group will receive repeated low-level red-light (R.L.R.L.) therapy twice daily using a no — Description:
  Participants in the experimental group will receive repeated low-level red-light (R.L.R.L.) therapy twice daily using a non-invasive light-emitting device. Each session will last no more than 3 minutes, with a minimum interval of 4 hours between sessions. The therapy is administered under parental supervision and aims to enhance myopia control in conjunction with orthokeratology.
  Arms: Experimental Arm Title: Orthokeratology + Red-Light Therapy Control Arm Title: Orthokeratology Only

SUMMARY:
This clinical trial investigates the efficacy of combining orthokeratology (OK) lenses with repeated low-level red-light (R.L.R.L.) therapy in slowing the progression of myopia in children classified as ortho-k non-responders. The MADRID study is a single-centre, prospective, randomized controlled trial conducted at the Centro Fernández-Velázquez in Madrid, Spain. Participants aged 8 to 15 years will be randomly assigned to either a control group (OK lenses only) or an experimental group (OK lenses + R.L.R.L. therapy). The primary objective is to assess the potential additive effect of R.L.R.L. therapy on axial length control over a 6 to 12-month follow-up period. All participants will undergo ocular biometry and posterior segment OCT at regular intervals. The study is fully self-funded by the institution and adheres to rigorous ethical and safety standards.

DETAILED DESCRIPTION:
Background and Rationale Myopia is a growing public health concern worldwide, especially among children, due to its progressive nature and association with severe ocular complications later in life. Orthokeratology (OK) lenses are one of the most effective non-pharmacological interventions for myopia control, reducing axial elongation by up to 63%. However, a subset of children, referred to as "ortho-k non-responders", continue to exhibit rapid axial elongation despite consistent use of OK lenses.

Repeated low-level red-light (R.L.R.L.) therapy is a novel, non-invasive intervention that has shown promise in reducing myopia progression. Preliminary studies suggest its mechanism may involve choroidal thickening, potentially complementing the effects of OK lenses. This study seeks to evaluate whether the combination of OK and R.L.R.L. offers additive benefits in myopia control for this specific population.

Study Design and Objectives This is a prospective, single-centre, randomized controlled clinical trial. The trial is being conducted at the Centro Fernández-Velázquez (Madrid, Spain) and aims to recruit 10 participants aged 8-15 years who meet specific inclusion criteria, including documented poor response to orthokeratology alone.

Participants will be randomized into two groups:

Experimental Group: OK lens + R.L.R.L. therapy (2 sessions/day, 3 minutes/session, minimum 4-hour interval) Control Group: OK lens only The primary endpoint is the change in axial length over 6 months, with the possibility of extending the intervention and monitoring for up to 12 months. Secondary endpoints include changes in refractive error, choroidal thickness, and treatment tolerance.

Measurements and Timeline Axial length will be measured using the Oculus Myopia Master. Posterior segment imaging will be performed with Topcon Maestro OCT. All evaluations are scheduled at baseline, 1 month, 3 months, and 6 months, and-if extended-at 9 and 12 months. All measurements will be performed between 9 a.m. and 11 a.m. to minimize diurnal variation.

Safety and Ethics All participants and/or their guardians will sign an informed consent prior to enrollment. The study adheres to the principles of the Declaration of Helsinki. A detailed adverse event management and reporting protocol is in place. All serious adverse events (SAEs) will be reported to the relevant ethical committees within 72 hours.

Funding and Conflicts of Interest This trial is fully self-funded by the Centro Fernández-Velázquez. The investigators declare no financial or personal conflicts of interest.

Conclusion This study will provide important preliminary evidence on the combined use of OK lenses and red-light therapy in managing progressive myopia in children who are non-responsive to orthokeratology alone. If effective, this combined approach could be incorporated into standard care protocols for high-risk paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 15 years. Intention to undergo orthokeratology (OK) lens treatment. Spherical equivalent refractive error between -1.00 and -4.00 diopters in either eye.

Astigmatism no greater than 1.50 D in either eye. Best corrected visual acuity (BCVA) of 25/25 or better in both eyes. Birth weight of at least 1500 g. Classified as ortho-k non-responders: continued OK use with persistent rapid myopia progression.

Willingness of child and legal guardian to participate and attend follow-up visits.

Signed informed consent by parent or guardian.

Exclusion Criteria:

* cular conditions such as strabismus, amblyopia, cataract, or ptosis. Previous use of OK lenses or atropine for myopia control. Contraindications to atropine (e.g., known allergy, cardiovascular disease, epilepsy).

Ocular contraindications to OK lens wear (e.g., inflammation, infection). Systemic diseases that may affect ocular growth (e.g., Down syndrome, Marfan syndrome).

Any other ocular disease that could interfere with study outcomes.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Axial Length | 12 months
  Axial length (in millimetres) will be measured using the Myopia Master (Oculus) at baseline and at 6 and 12 months to evaluate the progression of myopia. Measurements will be conducted between 9:00-11:00 a.m. to reduce diurnal variation.

SECONDARY OUTCOMES:
Change in Refractive Error (Spherical Equivalent) at 6 and 12 Months | 12 months
  Change in spherical equivalent refraction (in dioptres) from baseline to 6 and 12 months will be assessed via cycloplegic autorefraction and subjective refraction to monitor refractive progression.
Change in Subfoveal Choroidal Thickness at 6 and 12 Months | 12 months
  Subfoveal choroidal thickness will be measured using spectral-domain OCT (Topcon Maestro) at baseline, 6 months, and 12 months to assess structural retinal changes potentially associated with treatment efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Miopia Fernandez-Velazquez, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared for this study due to the small sample size, the exploratory nature of the investigation, and privacy considerations. Future larger-scale studies may consider data sharing under appropriate governance.

REFERENCES:
- [Background] Jiang Y, Zhu Z, Tan X, Kong X, Zhong H, Zhang J, Xiong R, Yuan Y, Zeng J, Morgan IG, He M. Effect of Repeated Low-Level Red-Light Therapy for Myopia Control in Children: A Multicenter Randomized Controlled Trial. Ophthalmology. 2022 May;129(5):509-519. doi: 10.1016/j.ophtha.2021.11.023. Epub 2021 Dec 1. PMID 34863776